CLINICAL TRIAL: NCT02530866
Title: Randomized Controlled Clinical Pilot Trial of Intensive Management for Gestational Diabetes
Brief Title: Intensive Management for Gestational Diabetes
Acronym: GDM-MOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5446
Record Dates: First submitted 2015-08-10; First posted 2015-08-21 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): Women in this arm will target fasting blood glucose values <95 mg/dL and 1 hour post-prandial values <140 mg/dL
  Interventions: Other: Lower glycemic targets
- Intensive therapy (Experimental): Women in the arm will target fasting blood glucose values <90 mg/dL and 1 hour post-prandial values <120 mg/dL.
  Interventions: Other: Lower glycemic targets

INTERVENTIONS:
Other: Lower glycemic targets — Women will be randomized to either standard or lower glycemic targets.

SUMMARY:
This is a randomized clinical pilot trial designed to assess the feasibility of randomizing obese women with GDM to lower glycemic thresholds compared to standard care. Maternal and cord blood metabolic profiles, neonatal body composition, and maternal sleep quality and duration will also be compared between groups.

DETAILED DESCRIPTION:
The investigators will randomize 60 obese pregnant women with a new diagnosis of gestational diabetes using the Carpenter-Coustan criteria in a 1:1 fashion to either standard care or intensive therapy. Subjects will be randomized to either standard care or intensive therapy at the first study visit, which will occur between 12-32 weeks of gestation after they have completed their gestational diabetes testing. Neither patients nor their providers will be blinded to patient study group. All women will receive standard nutritional counseling at the time of diagnosis, and they will also be treated with either glyburide or insulin as dictated by standard care. Women will return for a second study visit between 32-36 weeks of gestation to assess the impact of their glycemic target groups on overall glycemic control. The investigators will also collect information on the type and dose of each medication required to maintain glycemic control in women randomized to either standard care or intensive therapy.

In addition to standard glucose monitoring 4x/day (fasting and one-hour post breakfast, lunch, and dinner), the investigators will utilize blinded continuous glucose monitors (iPro, Medtronic) at each study visit. Because women with GDM are receiving active management of their blood sugars and dietary counseling, the investigators will assess CGM for 5 consecutive days both at study enrollment and again between 32-36 weeks. Study participants will complete food diaries during their CGM monitoring to correlate food intake with glycemic variation. The investigators will also compare maternal and cord blood metabolic profiles, neonatal body composition, and maternal sleep quality and duration between groups.

ELIGIBILITY:
Inclusion Criteria:

* maternal age between 18-45 years
* singleton birth
* planned delivery at OU Medical Center
* GDM diagnosed between 12-32 weeks' gestation by either a 50 gram
* one hour GCT >200 mg/dL or two or more abnormal values on a 100 gram OGTT using the Carpenter-Coustan criteria
* pre-pregnancy BMI ≥26 kg/m2.

Exclusion Criteria:

* maternal tobacco use
* planned delivery prior to 34 weeks of gestation
* significant fetal anomalies
* chronic hypertension requiring medication
* other vascular disease
* known renal disease with a baseline serum creatinine >1.5 mg/dL
* maternal rheumatologic disorders requiring medication
* maternal human immunodeficiency virus (HIV) or hepatitis
* as the specimen storage facility is not accredited to handle such samples
* steroid use within 7 days.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change in baseline maternal glycemia at 32-36 weeks gestation | 5 days at 2 separate times (1st study visit at 12-32 weeks, 2nd study visit at 32-36 weeks)
  Women will undergo CGM for 5 days at both the first study visit (12-32 weeks) and again at the second study visit (32-36 weeks). Our primary outcome between women randomized to either SC or IT will compare mean 24-hour blood glucose levels as assessed by continuous glucose monitor at the 2nd study visit, which will occur between 32-36 weeks of gestation. Investigators hypothesize that women randomized to the IT group will have a 10 mg/dL lower mean 24-hour glucose as assessed by continuous glucose monitor when compared to women in the SC group. Investigators will also assess the prevalence of maternal hypoglycemia by comparing the amount of time with maternal blood glucose values <60 mg/dL between groups.

SECONDARY OUTCOMES:
Neonatal body composition | At birth
  Total body composition will compared among infants of mothers randomized to either SC and IT using air-displacement plethysmography (ADP).
Cytokine measurements | 20-30 weeks of gestation and 32-36 weeks of gestation
  Maternal and cord blood levels
Physical activity | 9 months
  Investigators will utilize the Actiwatch Spectrum Pro (Phillips Healthcare, Pittsburgh, PA) for assessment of both sleep and physical activity in women . Subjects will wear this device on their wrist at baseline and again at the 32-36 week follow-up visit. The Actiwatch monitoring periods are designed to coincide with the periods of CGM monitoring.
Sleep assessments | 9 months
  Investigators will utilize the Actiwatch Spectrum Pro (Phillips Healthcare, Pittsburgh, PA) for assessment of both sleep and physical activity in women . Subjects will wear this device on their wrist at baseline and again at the 32-36 week follow-up visit. The Actiwatch monitoring periods are designed to coincide with the periods of CGM monitoring.
Patient questionnaires | 9 months
  In order to help investigators understand the personal factors that lead to better glycemic control, patients will complete questionnaires regarding issues such as sleep, exercise, views about weight gain, mood, and stress levels.
Lipid measurements | 20-30 weeks of gestation and 32-36 weeks of gestation
Glucose measurements | 20-30 weeks of gestation and 32-36 weeks of gestation
Lipid profile measurements | 20-30 weeks of gestation and 32-36 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Pierce, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Scifres CM, Mead-Harvey C, Nadeau H, Reid S, Pierce S, Feghali M, Myers D, Fields D, Stoner JA. Intensive glycemic control in gestational diabetes mellitus: a randomized controlled clinical feasibility trial. Am J Obstet Gynecol MFM. 2019 Nov;1(4):100050. doi: 10.1016/j.ajogmf.2019.100050. Epub 2019 Sep 27. PMID 33345840